CLINICAL TRIAL: NCT06780020
Title: Effects of Different Interventions Using Boxing, Taekwondo and Elastic Band Training on Body Composition and Physical Performance in Chilean Older Women
Brief Title: Boxing, Taekwondo and Elastic Band Training on Body Composition and Physical Performance in Older Women
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica del Maule (Other)
Collaborators: Universidad Católica del Maule (UCM, Chile) (Unknown)
Responsible Party: Principal Investigator, Pablo Valdés-Badilla, Principal Investigator, Universidad Católica del Maule
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 29-2022
Record Dates: First submitted 2025-01-03; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Older People; Sports; Martial Arts
Keywords: Aging; Physical Functional; sports combat

STUDY DESIGN:
Intervention Model Description: In this study there is a randomized controlled trial, repeated measures, double-blinded participants and evaluators, and a quantitative approach for three parallel groups: BOX group, TKD group and EBT group.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Taekwondo group (Experimental): The TKD program was non-contact exercises (main part), which were broken up into 10 min of fundamental positions and particular technical foundations with the upper body (blocks and strikes) and 20 min of lower body technical foundations (movement, positions, and kicks), performed individually and in pairs with and without the use of taekwondo impact pads and shields; also, specific choreographies or poomsae (Kibom Poomsae and Il Jang) were performed for 10 min. During the first two weeks of training, three sets of eight repetitions of specific upper and lower limb technical fundamentals were performed, with a two-minute rest between sets . Weeks 3 to 5 saw an increase in volume, to four sets of eight repetitions for specific technical fundamentals, with a two-minute rest between sets. The sets were maintained at four during weeks 6, while the number of repetitions was increased to 12. Finally, the rest period was reduced to 90 s between weeks 7 and 8, while maintaining th
  Interventions: Other: Effects of different interventions using taekwondo
- Boxing (Experimental): For the BOX program, non-contact exercises were performed, during the main part of the class participants learned basic guard position movements, execution of isolated punches, and punch combinations. Rope jumping techniques were taught, including the swinging and rope jumping movement, ending with mental performance stimulation exercises such as breathing techniques, visualization and mental rehearsal, goal setting, and self-talk. The specific elements of each class varied beyond the 4 weeks, with a progression from learning simple exercises and simple drills and "fundamentals" to learning more complex movements and combinations. During the first two weeks of training, three sets of eight repetitions of basic movements and isolated punching techniques were performed with a two-minute rest between sets. Weeks 3 to 5 saw an increase in volume, to four sets of eight repetitions incorporating the execution of punch combinations (3 to 4 punches), with a two-minute rest between s
  Interventions: Other: Effects of different interventions using boxing
- Elastic band (Experimental): The EBT program is based on previous studies that demonstrated that it is safe and effective for older people. Using the TheraBand® elastic band system (Hygenic Corporation, Akron, OH, USA), participants started with a 10 min warm-up with joint mobility and low-intensity aerobic exercises. The colors of the elastic bands (yellow, red, green, blue, black, silver, and gold), each corresponding to a specific tension range, were used to indicate the training loads. The OMNI Resistance Exercise Scale (OMNI-RES) was used to monitor resistance training intensity, which ranged from moderate to vigorous (5 to 8 points). Six upper limb muscle strength exercises were done (pull-up, pullback, shoulder abduction, biceps curl, triceps, forearm) and 6 for the lower limbs (leg press, ankle eversion, ankle dorsiflexion, knee extension, knee flexion, and hip flexion). The older women started with the lowest resistance (yellow color), achieving a 10-repetition maximum (10 RM) of an upper an
  Interventions: Other: Effects of different interventions using Elastic Band

INTERVENTIONS:
Other: Effects of different interventions using boxing — The programs were designed to consist of 8 weeks (16 sessions) with a warm-up consisting of joint mobility and low-intensity aerobic activities, a 40-minute core component BOX and a 10-minute cool-down with static flexibility exercises.
  Other Names: BOXING
  Arms: Boxing
Other: Effects of different interventions using taekwondo — The programs were designed to consist of 8 weeks (16 sessions) with a warm-up consisting of joint mobility and low-intensity aerobic activities, a 40-minute core component TKD and a 10-minute cool-down with static flexibility exercises.
  Other Names: Taekwondo
  Arms: Taekwondo group
Other: Effects of different interventions using Elastic Band — The programs were designed to consist of 8 weeks (16 sessions) with a warm-up consisting of joint mobility and low-intensity aerobic activities, a 40-minute core component Elastic Band and a 10-minute cool-down with static flexibility exercises.
  Other Names: Elastic Band
  Arms: Elastic band

SUMMARY:
The objective of this clinical trial is to compare the effect of three physical interventions (Taekwondo, Boxing, and Elastic Band Training) on body composition and physical performance in older Chilean women. The main questions this study aims to answer are:

How do Taekwondo, Boxing, and Elastic Band Training affect body composition (body fat percentage and fat-free mass)?

What improvements are observed in physical performance (grip strength, balance, flexibility, and cardiorespiratory fitness) with each intervention?

Researchers will compare the effects of these three interventions to determine which offers the greatest benefits for body composition and physical performance.

Participants will:

Perform Taekwondo, Boxing, or Elastic Band Training twice a week for 8 weeks. Be assessed for morphological and physical performance variables before and after the intervention period.

Participate in supervised training sessions at local sports centers. This study aims to provide solid evidence on the efficacy of different physical interventions in improving the physical health of older women, helping to define more effective and accessible training strategies.

DETAILED DESCRIPTION:
Study Design In this study there is a randomized controlled trial, repeated measures, double-blinded participants and evaluators, and a quantitative approach for three parallel groups: BOX group, TKD group and EBT group. The randomization process was performed using the research randomizer website (https://www.randomizer.org, accessed March 1, 2023). CONSORT standards were used as the methodology. In addition, the protocol has been registered in ClinicalTrials.gov in the United States (code: ). The duration of the interventions was 8 weeks (16 sessions), including two weekly sessions on Tuesdays and Thursdays of sixty minutes each. Morphological variables (BMI, body fat percentage and fat-free mass), and functional performance, MIHS dominant and non-dominant hand, 30-second chair stand, TUG, sit and reach, back scratch and 2-minute walk were evaluated. Each measurement was performed at the same place (sports center and social headquarters) and in the afternoon, from 14:00 to 16:00, with the factors under control, including temperature, and the evaluators performing the pre- and post-measurements. With no musculoskeletal and/or cardiorespiratory injuries during the intervention, the older women showed no pain before the evaluations or during the training sessions.

Participants Sixty-three older women participated in the intervention at first. The optimal number of participants per group, according to the sample size calculation, was 10. Statistical power was calculated with the program GPower (version 3.1.9.6, Franz Faul, UniversiätKiel, Kiel, Germany). According to a previous study, the minimum difference necessary for significant clinical relevance was determined to be a mean difference of 0.50 s in the TUG, with a standarddeviation of 0.93 s, taking into account an alpha level of 0.05 with a power of 95% and a predicted loss of 10%. The inclusion requirements were: (i) women between 60 and 65 years of age; (ii) who demonstrated the ability to understand and execute instructions in a contextualized manner through basic directives; (iii) who were independent, according to a score of at least 43 points on the Chilean Ministry of Health's Preventive Medicine Examination for Older Adults; and (iv) who met the requirement of attendance at the intervention of at least 85%. In relation to the exclusion criteria, the following were taken into account (i) having a disability; (ii) undergoing physical rehabilitation or having musculoskeletal injuries that prevent them from performing their usual physical activities; and (iii) being permanently or temporarily unable to participate in physical activities. As for exclusion criteria, the following were taken into account: (i) suffering from a disability of any type; (ii) suffering from a musculoskeletal injury or receiving physical rehabilitation therapy that prevents them from performing their usual physical activity; and (iii) being unable to perform physical activity, either temporarily or permanently. To be included in the final analysis, participants who met the inclusion criteria also had to complete at least 85% of the training sessions and attend all evaluation sessions. The inclusion criteria are summarized in Figure 1.

ELIGIBILITY:
Inclusion Criteria:

* women between 60 and 65 years of age
* who demonstrated the ability to understand and execute instructions in a contextualized manner through basic directives
* who were independent, according to a score of at least 43 points on the Chilean Ministry of Health's Preventive Medicine Examination for Older Adults
* who met the requirement of attendance at the intervention of at least 85%.

Exclusion Criteria:

* having a disability
* undergoing physical rehabilitation or having musculoskeletal injuries that prevent them from performing their usual physical activities.
* being permanently or temporarily unable to participate in physical activities.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-04-04 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Bipedal height | 8 weeks
  Bipedal height was measured using a stadiometer (Seca model 220, SECA, Hamburg,Germany; accuracy to 0.1 cm).
Body weight | 8 weeks
  body weight was calculated using a mechanical scale(Scale-tronix, Chicago, IL, USA; accuracy to 0.1 kg) while wearing the barest minimum of clothing.
Thirty-Second Chair Stand (30-s chair stand) | 8 weeks
  The 30-s chair stand test counts the number of repetitions performed while sitting on the chair, with arms resting on the chest, for thirty seconds. It was designed to assess the muscular strength of the lower limbs. After three attempts with a recovery of 120 s between each, the best of the three efforts was attained.
Timed Up-and-Go (TUG) | 8 weeks
  The TUG test was carried out in accordance with previous recommendations. The person must get out of an arm-supported chair, travel a 3-m hallway, turn around, and return to the chair. They must swiftly record the best of three trials after completing them. Two assessors recorded the time using single-beam photocells (Brower Timing System, Draper, UT, USA); the best three attempts were statistically analyzed.
Sit-and-Reach Test | 8 weeks
  Utilizing the sit-and-reach test, flexibility was assessed. Subjects were seated forward in a chair with a fixed back, one leg bent on the floor and the other left straight. The left or right leg may be used to run comfortably; however, the post-test measured the same leg as the pre-test. After correcting the position once again, the case of another bent leg evaluates flexibility by executing two attempts using the higher number to determine the result.
Back scratch | 8 weeks
  For the Back Scratch Test, the participant placed one hand on the shoulder and one hand towards the middle of the back maintaining the position. The evaluator measured the amount of cm (+ or -) between the extended ring fingers of both hands.
2-min Step Test | 8 weeks
  Cardiorespiratory fitness was measured using the 2-min step test. Participants were instructed to stand straight, and the middle distance between the patella and pelvic bones was marked on a wall with colored tape. Participants stepped in a manner where their knees were raised above the marked spot, and the number of repetitions within 2 min was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Valdes-Badilla, Doctor, Principal Investigator — Universidad Cátolica del Maule
Locations (1):
- Universidad Católica del Maule, Talca, Maule Region, Chile

IPD SHARING:
Plan to Share IPD: No
The data will remain with the research team; due to the type of project, it cannot be shared.